CLINICAL TRIAL: NCT02137239
Title: Evaluation of Acute Rejection Rates in de Novo Renal Transplant Recipients Following Thymoglobulin Induction, CNI-free, Nulojix (Belatacept)-Based Immunosuppression
Brief Title: Regimen Optimization Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IM103-177; 2013-002090-21 (EudraCT Number)
Record Dates: First submitted 2014-05-12; First posted 2014-05-13 (Estimated); Results first posted 2021-06-22 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-05

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — thymoglobulin; Abatacept; Mycophenolic Acid; Adrenal Cortex Hormones; Methylprednisolone; Prednisone; Everolimus; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Belatacept + Everolimus (Experimental): Thymoglobulin (i.v. infusion) induction, daily (or less frequently, as tolerated) not to exceed 10 days, to reach a total cumulative dose between 3.0 and 5.5 mg/kg; belatacept (infusion) regimen of 10 mg/kg i.v. on Day 1, Weeks 1, 2, 4, 8 and 12 post transplant and then a maintenance dose of 5 mg/kg every 4 weeks after 12 weeks post transplant; everolimus (tablet) daily dosing at 3.0 mg/day, 2 divided doses, starting on Day 3 dosing adjusted based on blood sample tests; methylprednisolone (infusion) prior to each Thymoglobulin infusion and prednisone (tablet), once methylprednisolone is no longer needed. (Corticosteroids to be discontinued by Day 7 or as soon thereafter as thymoglobulin infusions are completed)
  Interventions: Drug: Thymoglobulin; Drug: Belatacept; Drug: Corticosteroids; Drug: Everolimus(EVL)
- Tacrolimus + Mycophenolate mofetil (Experimental): Thymoglobulin (i.v. infusion) induction, daily (or less frequently, as tolerated) not to exceed 10 days, to reach a total cumulative dose between 3.0 and 5.5 mg/kg; tacrolimus (tablet) daily dosing beginning at 0.1 mg/kg/day, then adjusted based on blood sample tests; MMF (tablet) daily dosing between 0.5 to 2.0 g/day divided in 2 doses (up to 3 g/day if African Americans/Blacks); methylprednisolone (infusion) prior to each Thymoglobulin infusion and prednisone (tablet), once methylprednisolone is no longer needed. (Corticosteroids to be discontinued by Day 7 or as soon thereafter as thymoglobulin infusions are completed)
  Interventions: Drug: Thymoglobulin; Drug: mycophenolate mofetil(MMF); Drug: Corticosteroids; Drug: Tacrolimus(TAC)

INTERVENTIONS:
Drug: Thymoglobulin
  Other Names: ATG
Drug: Belatacept
  Other Names: Nulojix
  Arms: Belatacept + Everolimus
Drug: mycophenolate mofetil(MMF)
  Other Names: CellCept
  Arms: Tacrolimus + Mycophenolate mofetil
Drug: Corticosteroids
  Other Names: Methylprednisolone; Prednisone
Drug: Everolimus(EVL)
  Other Names: Certican®; Zortress®
  Arms: Belatacept + Everolimus
Drug: Tacrolimus(TAC)
  Other Names: Prograf
  Arms: Tacrolimus + Mycophenolate mofetil

SUMMARY:
Patients who undergo a kidney transplant require prolonged therapy with drugs that suppress the immune system (called immunosuppressive regimens) to stop the immune system from attacking the transplanted kidney in order to limit damage to or the possibility of rejecting the transplanted kidney. The purpose of this study is to evaluate benefits and risks of two immunosuppressive regimens (belatacept with everolimus or tacrolimus with mycophenolate mofetil) following thymoglobulin induction and rapid corticosteroid withdrawal.

DETAILED DESCRIPTION:
Calcineurin inhibitor (CNI)

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Men and women, aged 18 to 75
* Serologic test results are positive for past exposure to Epstein Barr Virus (EBV+)
* Diagnosed with end stage renal disease (ESRD) and scheduled to undergo transplantation of a non-HLA identical, living or standard criteria deceased donor kidney

Exclusion Criteria:

* Primary cause of ESRD is: primary focal segmental glomerulosclerosis; or Type I or II membranoproliferative glomerulonephritis; or Hemolytic Uremic Syndrome / Thrombotic Thrombocytopenic Purpura
* Had a previous graft loss due to acute rejection
* At increased immunologic risk of graft loss due to panel reactive antibodies (PRA) >20% or need for desensitization therapy
* Scheduled to receive a: kidney from identical twin; or paired kidney; or kidney from a Cytomegalovirus(CMV) positive donor when recipient is CMV negative; or kidney from an extended criteria donor
* Have a body mass index (BMI) of > 35 kg/m2 for nondiabetics or > 30 kg/m2 for diabetics
* Diagnosed as Hepatitis B positive; or Hepatitis C positive; or HIV positive; or currently or previously active or inadequately treated latent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2015-12-31 (Actual); Primary Completion 2019-05-02 (Actual); Study Completion 2019-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (20):
- United States (17):
  - California Institute Of Renal Research, San Diego, California
  - California Pacific Medical Center, San Francisco, California
  - University Of Colorado, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Emory Univeristy, Atlanta, Georgia
  - University Of Illinois, Chicago, Illinois
  - Tulane Medical Center, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Erie County Medical Center, Buffalo, New York
  - Wake Forest University School Of Medicine, Winston-Salem, North Carolina
  - Central PA Transplant Foundation, Harrisburg, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Virginia, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Swedish Medical Center - Swedish Colon and Rectal Clinic - First Hill (Northwest Colon and Rectal Cl, Seattle, Washington
- Argentina (3):
  - Sanatorio Parque S.A., Rosario, Santa Fe Province
  - Clinica Privada Velez Sarsfield, Córdoba
  - Clinica De Nefrologia, Urologia Y Enf. Cardiovasculares, Sante Fe

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 58 participants randomized and treated
Groups:
- Treatment A: BELA + EVL
- Treatment B: TAC + MMF
Period: Overall Study
Arm/Group | Treatment A | Treatment B
Started | 26 | 32
Completed | 23 | 26
Not Completed | 3 | 6
Not completed — Discontinued Study Treatment | 0 | 3
Not completed — Withdrew Consent | 1 | 1
Not completed — Adverse Event | 2 | 2

BASELINE CHARACTERISTICS:
Population: Randomized, Transplanted and Treated Population (ITT)
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment A | Treatment B | Total
Number analyzed (Participants) | 26 | 32 | 58
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.7 (12.8) | 50.8 (10.9) | 51.2 (11.7)
Age, Customized [Count of Participants; unit: Participants]
  < 65 | 22 | 28 | 50
  ≥ 65 | 4 | 4 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 14
  Male | 21 | 23 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 6 | 9
  White | 23 | 21 | 44
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Clinically-suspected Biopsy-proven Acute Rejection (CSBPAR) at 6 Months
Description: Number of Participants with Clinically-suspected biopsy-proven acute rejection (CSBPAR) at 6 Months
Time Frame: 6 Months
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 26 | 32
Percentage of participants | 7.7 [0.9 to 25.1] | 9.4 [2.0 to 25.0]

2. Secondary Outcome: Clinically-suspected Biopsy-proven Acute Rejection (CSBPAR) at 6, 12 and 24 Months
Description: Clinically-suspected biopsy-proven acute rejection (CSBPAR) at 6, 12 and 24 Months
  Change in the incidence of CSBPAR at 6, 12 and 24 months post transplant, in the belatacept + EVL(Treatment A) as compared to TAC + MMF (Treatment B).
Time Frame: Up to 24 Months
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: Percentage of CSBPAR
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 26 | 32
Percentage of CSBPAR
  CSBPAR at 6 Months | 7.7 [0.9 to 25.1] | 9.4 [2.0 to 25.0]
  CSBPAR at 12 months | 11.5 [2.4 to 30.2] | 12.5 [3.5 to 29.0]
  CSBPAR at 24 Months | 15.4 [4.4 to 34.9] | 12.5 [3.5 to 29.0]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Change in Incidence of Treatment A as compared to Treatment B at 6 Months; Test type: Superiority; Incidence of Change = -1.7, 95% CI 2-sided [-18.9 to 16.7]
Statistical Analysis 2: Comparison: Treatment A vs Treatment B; Change in Incidence of Treatment A as compared to Treatment B at 12 Months; Test type: Superiority; Incidence of Change = -1.0, 95% CI 2-sided [-19.2 to 18.9]
Statistical Analysis 3: Comparison: Treatment A vs Treatment B; Change in Incidence of Treatment A as compared to Treatment B at 24 Months; Test type: Superiority; Incidence of Change = 2.9, 95% CI 2-sided [-16.1 to 23.9]

3. Secondary Outcome: Time to Clinically-suspected Biopsy-proven Acute Rejection (CSBPAR).
Description: Time to Clinically suspected biopsy proven acute rejection
Time Frame: Up to 24 Months
Population: Participants with a CSBPAR
Measure: Mean (Full Range); unit: Months
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 3 | 3
Months | NA [NA to NA] — Randomization Error: See limitations and caveats | NA [NA to NA] — Randomization Error: See limitations and caveats

4. Secondary Outcome: Percentage of Participants With BANFF Grade by Severity Grades. BANFF Type (Grade) for Acute/Active Rejection
Description: Treatment differences in the severity grades to treat all episodes of CSBPAR at 6, 12, and 24 months post-transplant.
  Type 1A - Cases with significant interstitial infiltration (>25% of parenchyma affected) and foci of moderate tubulitis (>4 mononuclear cells/Tubular cross section or group of 10 Tubular cell). Type 1B - Cases with significant interstitial infiltration (>25% of parenchyma affected) and foci of moderate tubulitis (>10 mononuclear cells/Tubular cross section or group of 10 Tubular cell).Type 2A - Cases with mild to moderate intimal arteritis.Type 2B - Cases with severe intimal arteritis comprising >25% of the luminal area. Type 3 - Cases with "transmural" arteritis and/or arterial fibrinoid change and necrosis of medial smooth muscle cells (v3 with accompanying lymphocytic inflammation)
Time Frame: At 6, 12 and 24 Months
Population: ITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 26 | 32
Percentage of Participants
  6 Months: Mild Acute (1A) | 3.8 | 0
  6 Months: Mild Acute (1B) | 0 | 3.1
  6 Months: Moderate Acute (2A) | 7.7 | 6.3
  6 Months: Moderate Acute (2B) | 0 | 0
  6 Months: Severe Acute | 0 | 0
  12 Months: Mild Acute (1A) | 7.7 | 3.1
  12 Months: Mild Acute (1B) | 0 | 3.1
  12 Months: Moderate Acute (2A) | 7.7 | 6.3
  12 Months: Moderate Acute (2B) | 0 | 0
  12 Months: Severe Acute | 0 | 0
  24 Months: Mild Acute (1A) | 11.5 | 3.1
  24 Months: Mild Acute (1B) | 0 | 3.1
  24 Months: Moderate Acute (2A) | 7.7 | 6.3
  24 Months: Moderate Acute (2B) | 0 | 0
  24 Months: Severe Acute | 0 | 0

5. Secondary Outcome: Treatment Differences in Therapeutic Modalities
Description: Treatment Received for Biopsy Proven Acute Rejection (Banff Grade IA or Higher), or Humoral (Antibody Mediated) Rejection Treatment regimen: Categorical analysis of CSBPAR episodes by treatment received.
Time Frame: at 6, 12 and 24 Months
Population: All Randomized, Transplanted and Treated Participants
Measure: Number; unit: Percentage of participants with CSBPARs
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 26 | 32
Percentage of participants with CSBPARs
  Corticosteroids (6 months) | 7.7 | 9.4
  Lymphocyte depleting agent (6 months) | 0 | 6.3
  Plasmapheresis (6 months) | 0 | 0
  IVIG (6 months) | 0 | 3.1
  Rituximab (6 months) | 0 | 0
  Corticosteroids (12 months) | 15.4 | 12.5
  Lymphocyte depleting agent (12 months) | 3.8 | 6.3
  Plasmapheresis (12 months) | 0 | 0
  IVIG (12 months) | 0 | 3.1
  Rituximab (12 months) | 0 | 0
  Corticosteroids (24 months) | 19.2 | 12.5
  Lymphocyte depleting agent (24 months) | 3.8 | 6.3
  Plasmapheresis (24 months) | 0 | 0
  IVIG (24 months) | 0 | 3.1
  Rituximab (24 months) | 0 | 0

6. Secondary Outcome: Number of Participants Who Survive With a Functioning Graft
Description: Number of all participants who survive with a functioning graft at 6, 12 and 24 months post transplant
Time Frame: At 6, 12 and 24 months
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 26 | 32
Participants
  At 6 Months | 25 | 31
  At 12 Months | 25 | 31
  At 24 Months | 25 | 31

7. Secondary Outcome: Number of Participants Deaths Post Transplant
Description: Number of participant deaths at 6, 12 and 24 months post transplant
Time Frame: up to 24 months
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 26 | 32
Participants
  At 6 Months | 0 | 0
  At 12 Months | 0 | 0
  At 24 Months | 0 | 0

8. Secondary Outcome: Number of Participants Who Experience Graft Loss Post Transplant
Description: Number of all participants who experience graft loss at 6, 12 and 24 months post transplant
Time Frame: At 6, 12 and 24 months
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 26 | 32
Participants
  At 6 Months | 1 | 1
  At 12 Months | 1 | 1
  At 24 Months | 1 | 1

9. Secondary Outcome: Time to Event: Graft Loss and Death
Description: The Number of days to participant Graft Loss and death for any reason
Time Frame: Up to 728 Days
Population: All Treated Participants
Measure: Number; unit: Days
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 1 | 1
Days
  Graft Loss | 107 | 2
  Death: number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Absolute Calculated Glomerular Filtration Rate (cGFR): Mean
Description: Absolute (mean and median) cGFR values at 3, 6, 12 and 24 months post-transplant, as determined from the 4-variable Modification of Diet in Renal Disease (MDRD) formula
Time Frame: Up 24 Months post-transplant
Population: ITT Population
Measure: Mean (95% Confidence Interval); unit: mL/min/1.73 m^2
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 26 | 32
mL/min/1.73 m^2
  At 3 Months: number analyzed (Participants) | 25 | 31
  At 3 Months | 69.2 [60.2 to 78.3] | 62.2 [55.3 to 69.1]
  At 6 Months: number analyzed (Participants) | 25 | 31
  At 6 Months | 66.0 [55.8 to 76.2] | 63.9 [56.2 to 71.5]
  At 12 Months: number analyzed (Participants) | 25 | 31
  At 12 Months | 66.2 [56.9 to 75.4] | 62.0 [53.4 to 70.6]
  At 24 Months: number analyzed (Participants) | 24 | 25
  At 24 Months | 71.8 [62.5 to 81.0] | 68.7 [59.2 to 78.2]

11. Secondary Outcome: Median Calculated Glomerular Filtration Rate (cGFR)
Description: Median cGFR values at 3, 6, 12 and 24 months post-transplant, as determined from the 4-variable Modification of Diet in Renal Disease (MDRD) formula
Time Frame: Up 24 Months post-transplant
Population: ITT Population
Measure: Median (Full Range); unit: mL/min/1.73 m^2
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 26 | 32
mL/min/1.73 m^2
  At 3 Months: number analyzed (Participants) | 25 | 31
  At 3 Months | 64.0 [52.0 to 80.0] | 62.0 [55.0 to 79.0]
  At 6 Months: number analyzed (Participants) | 25 | 31
  At 6 Months | 64.0 [56.0 to 79.0] | 67.0 [55.0 to 75.0]
  At 12 Months: number analyzed (Participants) | 25 | 31
  At 12 Months | 66.0 [58.0 to 77.0] | 62.5 [47.5 to 74.0]
  At 24 Months: number analyzed (Participants) | 24 | 25
  At 24 Months | 73.5 [59.5 to 84.5] | 68.0 [56.0 to 82.0]

12. Secondary Outcome: Mean Change From Month 3 in cGFR
Description: The mean change from Month 3 cGFR at 3, 6, 12 and 24 months post-transplant
Time Frame: Up 24 Months post-transplant
Population: ITT Population
Measure: Mean (95% Confidence Interval); unit: mL/min/1.73 m^2
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 26 | 32
mL/min/1.73 m^2
  At 3 Months: number analyzed (Participants) | 25 | 31
  At 3 Months | 0 [0 to 0] | 0 [0 to 0]
  At 6 Months: number analyzed (Participants) | 25 | 31
  At 6 Months | -3.2 [-10.9 to 4.5] | 2.8 [-0.2 to 5.8]
  At 12 Months: number analyzed (Participants) | 25 | 31
  At 12 Months | -3.1 [-12.6 to 6.5] | 1.4 [-3.3 to 6.0]
  At 24 Months: number analyzed (Participants) | 24 | 25
  At 24 Months | 3.1 [-4.2 to 10.4] | 6.3 [-0.6 to 13.2]

13. Secondary Outcome: Urine Protein Creatinine Ratio (UPr/Cr)
Description: Urine protein to creatinine ratio (UPr/Cr) at 3, 6, 12 and 24 months post-transplant.
Time Frame: Up 24 Months post-transplant
Population: ITT Population
Measure: Mean (95% Confidence Interval); unit: mg Protein/mg Creatinine
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 26 | 32
mg Protein/mg Creatinine
  At 3 Months: number analyzed (Participants) | 25 | 27
  At 3 Months | 0.3146 [0.1985 to 0.4307] | 0.1412 [0.1097 to 0.1726]
  At 6 Months: number analyzed (Participants) | 25 | 27
  At 6 Months | 0.3896 [0.2326 to 0.5466] | 0.1461 [0.1203 to 0.1720]
  At 12 Months: number analyzed (Participants) | 23 | 24
  At 12 Months | 0.2835 [0.1648 to 0.4021] | 0.1849 [0.1041 to 0.2658]
  At 24 Months: number analyzed (Participants) | 20 | 23
  At 24 Months | 0.3940 [0.2199 to 0.5680] | 0.1685 [0.1174 to 0.2195]

14. Secondary Outcome: Percentage of Participants With Donor Specific Anti-HLA Antibodies (DSA)
Description: Percentage of participants with, and titers of pre-existing (pre-transplant) DSA on Day 1 (pre-transplant, pre-dose), and at Months 12 and 24 posttransplant
Time Frame: Up to 24 Months
Population: As Treated Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 25 | 33
Percentage of Participants
  Baseline Class 1 DSA: number analyzed (Participants) | 20 | 29
  Baseline Class 1 DSA | 10 | 0
  Baseline Class 2 DSA: number analyzed (Participants) | 20 | 29
  Baseline Class 2 DSA | 0 | 0
  Baseline Both Class 1 and 2 DSA: number analyzed (Participants) | 20 | 29
  Baseline Both Class 1 and 2 DSA | 0 | 0
  12 Month Class 1 DSA | 8.00 | 0
  12 Month Class 2 DSA | 0 | 3.03
  12 Month Both Class 1 and 2 DSA | 0 | 0
  24 Month Class 1 DSA | 8.00 | 3.03
  24 Month Class 2 DSA | 0 | 3.03
  24 Month Both Class 1 and 2 DSA | 0 | 0

15. Secondary Outcome: Percentage of Participants With De Novo Donor Specific Anti-HLA Antibodies (DSA)
Description: Characterization of any de novo DSA detected by IgM and IgG subclasses, and by the presence or absence of complement fixing properties.
Time Frame: Up to 24 Months
Population: As Treated Population
Measure: Number; unit: Percentage
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 25 | 33
Percentage
  Baseline Class 1 DSA: number analyzed (Participants) | 20 | 29
  Baseline Class 1 DSA | 10 | 0
  Baseline Class 2 DSA: number analyzed (Participants) | 20 | 29
  Baseline Class 2 DSA | 0 | 0
  Baseline Both Class 1 and 2 DSA: number analyzed (Participants) | 20 | 29
  Baseline Both Class 1 and 2 DSA | 0 | 0
  De Novo 12 Month Class 1 DSA: number analyzed (Participants) | 25 | 29
  De Novo 12 Month Class 1 DSA | 0 | 0
  De Novo 12 Month Class 2 DSA: number analyzed (Participants) | 25 | 29
  De Novo 12 Month Class 2 DSA | 0 | 0
  De Novo 12 Month Both Class 1 and 2 DSA: number analyzed (Participants) | 25 | 29
  De Novo 12 Month Both Class 1 and 2 DSA | 0 | 0
  De Novo 24 Month Class 1 DSA: number analyzed (Participants) | 20 | 29
  De Novo 24 Month Class 1 DSA | 0 | 3.45
  De Novo 24 Month Class 2 DSA: number analyzed (Participants) | 20 | 29
  De Novo 24 Month Class 2 DSA | 0 | 0
  De Novo 24 Month Both Class 1 and 2 DSA: number analyzed (Participants) | 20 | 29
  De Novo 24 Month Both Class 1 and 2 DSA | 0 | 0

16. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: Percentage of participants with AEs up to 24 months post-transplant
Time Frame: Up to 24 months Post-Transplant
Population: As Treated Population
Measure: Number; unit: Percentage of participants with AEs
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 25 | 33
Percentage of participants with AEs | 100.0 | 97.0

17. Secondary Outcome: Percentage of Participants With Serious Adverse Events (SAEs)
Description: Percentage of participants with SAEs up to 24 months post-transplant
Time Frame: Up to 24 months Post-Transplant
Population: As Treated Population
Measure: Number; unit: Percentage of participants with SAEs
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 25 | 33
Percentage of participants with SAEs | 52.0 | 60.6

18. Secondary Outcome: Percentage of Participants With Events of Special Interest (ESIs)
Description: Percentage of participants which have one of the following events of special interest:
  Serious Infections Post-Transplant Lymphoproliferative Disorder (PTLD) Progressive multifocal leukoencephalopathy (PML) Malignancies (Other than PTLD) including non-melanoma skin carcinomas (Malignancies) Tuberculosis Infections Central Nervous System (CNS) Infections Viral Infections Infusion Related reactions within 24 hours since belatacept infusion
Time Frame: Up to 24 Months
Population: As Treated Population
Measure: Number; unit: Percentage of participants with ESIs
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 25 | 33
Percentage of participants with ESIs
  Serious Infections | 16 | 15.2
  PTLD | 4.0 | 3.0
  PML | 0 | 0
  Malignancies | 4.0 | 3.0
  TB | 0 | 0
  CNS Infections | 0 | 0
  Viral Infections | 0 | 0
  Infusion Related Reactions | 1 | 0

19. Secondary Outcome: Percentage of Particpants With Laboratory Test Abnormalities (LTAs)
Description: Percentage of participants with laboratory tests with marked laboratory abnormalities
Time Frame: At 24 Months
Population: As Treated Population
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 25 | 33
Percentage of participants
  Hemoglobin (Low) | 12.0 | 6.1
  Leukocytes (low) | 0 | 3.0
  Lymphocyte (Absolute) (low) | 84.0 | 69.7
  Neutrophils (Absolute) (low) | 0 | 3.0
  Aspartate Aminotransferase (High) | 4.0 | 0
  Creatinine (High) | 16.0 | 3.0
  Inorganic Phosphorus (low) | 24.0 | 12.1
  Potassium (high) | 4.0 | 0
  Sodium (low) | 4.0 | 0
  Albumin (low) | 0 | 3.0
  Glucose (high) | 8.0 | 12.1
  Triglycerides (high) | 12.0 | 0
  Uric Acid (high) | 8.0 | 0

20. Secondary Outcome: Mean and Mean Change From Baseline in Blood Glucose
Description: Mean fasting blood glucose levels, and mean changes from baseline values at Months 6, 12 and 24 months post- transplant
Time Frame: Up to 24 months
Population: ITT Population
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 26 | 32
mg/dL
  Mean Value at 6 months: number analyzed (Participants) | 20 | 25
  Mean Value at 6 months | 107.2 [86.6 to 127.8] | 107.2 [93.8 to 120.7]
  Change from baseline at 6 months: number analyzed (Participants) | 18 | 20
  Change from baseline at 6 months | 4.9 [-5.8 to 15.7] | 4.8 [-17.6 to 27.2]
  Mean Value at 12 months: number analyzed (Participants) | 23 | 24
  Mean Value at 12 months | 101.1 [85.3 to 117.0] | 127.5 [99.2 to 155.8]
  Change from baseline at 12 months: number analyzed (Participants) | 20 | 18
  Change from baseline at 12 months | -1.3 [-24.7 to 22.1] | 20.6 [0.4 to 40.8]
  Mean Value at 24 months: number analyzed (Participants) | 17 | 19
  Mean Value at 24 months | 127.5 [93.7 to 161.4] | 111.8 [87.1 to 136.5]
  Change from baseline at 24 months: number analyzed (Participants) | 14 | 14
  Change from baseline at 24 months | 22.3 [-15.7 to 60.3] | 15.0 [-3.2 to 33.2]

21. Secondary Outcome: Mean and Mean Change From Baseline in Whole Blood HbA1c
Description: Mean whole blood HbA1C concentrations, and mean changes from baseline values at Months 6, 12 and 24 months post-transplant.
Time Frame: Up to 24 months
Population: ITT Population
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 26 | 32
mg/dL
  Mean Value at 6 months: number analyzed (Participants) | 22 | 26
  Mean Value at 6 months | 6.11 [5.47 to 6.75] | 6.13 [5.44 to 6.82]
  Change from baseline at 6 months: number analyzed (Participants) | 22 | 25
  Change from baseline at 6 months | 0.34 [0.06 to 0.62] | 0.48 [0.04 to 0.91]
  Mean Value at 12 months: number analyzed (Participants) | 24 | 24
  Mean Value at 12 months | 6.18 [5.42 to 6.93] | 6.21 [5.50 to 6.92]
  Change from baseline at 12 months: number analyzed (Participants) | 23 | 23
  Change from baseline at 12 months | 0.47 [-0.00 to 0.95] | 0.32 [-0.17 to 0.81]
  Mean Value at 24 months: number analyzed (Participants) | 19 | 22
  Mean Value at 24 months | 6.24 [5.27 to 7.20] | 6.29 [5.38 to 7.20]
  Change from baseline at 24 months: number analyzed (Participants) | 18 | 21
  Change from baseline at 24 months | 0.66 [-0.05 to 1.37] | 0.41 [-0.13 to 0.95]

22. Secondary Outcome: Percentage of Participants With New Onset Diabetes After Transplant
Description: Percentage of participants with New Onset Diabetes After Transplantation (NODAT) at 6, 12, and 24 months post-transplant.
Time Frame: up to 24 months
Population: ITT Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 26 | 32
Percentage of participants
  Up to 6 Months | 11.5 [2.4 to 30.2] | 6.3 [0.8 to 20.8]
  Up to 12 Months | 11.5 [2.4 to 30.2] | 6.3 [0.8 to 20.8]
  Up to 24 Months | 15.4 [4.4 to 34.9] | 12.5 [3.5 to 29.0]

23. Secondary Outcome: Absolute Values of Blood Pressure: Mean
Description: Absolute (mean and median) values for SBP and DBP at 3, 6, 12 and 24 months posttransplant;
Time Frame: Up to 24 Months
Population: ITT Population
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 26 | 32
mmHg
  Diastolic Month 3: number analyzed (Participants) | 26 | 30
  Diastolic Month 3 | 78.7 [74.2 to 83.2] | 77.7 [74.0 to 81.3]
  Systolic Month 3: number analyzed (Participants) | 26 | 30
  Systolic Month 3 | 134.2 [126.9 to 141.6] | 131.0 [124.9 to 137.0]
  Diastolic Month 6: number analyzed (Participants) | 24 | 28
  Diastolic Month 6 | 77.4 [73.6 to 81.3] | 79.4 [76.0 to 82.9]
  Systolic Month 6: number analyzed (Participants) | 24 | 28
  Systolic Month 6 | 128.1 [121.8 to 134.5] | 133.0 [127.2 to 138.8]
  Diastolic Month 12: number analyzed (Participants) | 24 | 27
  Diastolic Month 12 | 78.7 [74.6 to 82.9] | 80.1 [76.4 to 83.8]
  Systolic Month 12: number analyzed (Participants) | 24 | 27
  Systolic Month 12 | 131.0 [125.6 to 136.4] | 131.0 [123.4 to 138.7]
  Diastolic Month 24: number analyzed (Participants) | 23 | 24
  Diastolic Month 24 | 78.1 [74.2 to 81.9] | 78.5 [74.3 to 82.8]
  Systolic Month 24: number analyzed (Participants) | 23 | 24
  Systolic Month 24 | 130.9 [125.2 to 136.5] | 131.7 [125.2 to 138.2]

24. Secondary Outcome: Absolute Values of Blood Pressure: Median
Description: Absolute (mean and median) values for SBP and DBP at 3, 6, 12 and 24 months posttransplant;
Time Frame: Up to 24 Months
Population: ITT Population
Measure: Median (Full Range); unit: mmHg
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 26 | 32
mmHg
  Diastolic Month 3: number analyzed (Participants) | 26 | 30
  Diastolic Month 3 | 78.5 [70.0 to 88.0] | 80.0 [70.0 to 84.0]
  Systolic Month 3: number analyzed (Participants) | 26 | 30
  Systolic Month 3 | 135.5 [127.0 to 144.0] | 131.0 [122.0 to 138.0]
  Diastolic Month 6: number analyzed (Participants) | 24 | 28
  Diastolic Month 6 | 75.5 [70.5 to 83.0] | 80.0 [71.0 to 85.5]
  Systolic Month 6: number analyzed (Participants) | 24 | 28
  Systolic Month 6 | 127.0 [114.5 to 136.5] | 131.0 [124.0 to 142.5]
  Diastolic Month 12: number analyzed (Participants) | 24 | 27
  Diastolic Month 12 | 77.0 [71.5 to 86.0] | 81.0 [72.0 to 88.0]
  Systolic Month 12: number analyzed (Participants) | 24 | 27
  Systolic Month 12 | 130.0 [119.0 to 142.0] | 126.0 [115.0 to 146.0]
  Diastolic Month 24: number analyzed (Participants) | 23 | 24
  Diastolic Month 24 | 78.0 [71.0 to 86.0] | 79.0 [69.5 to 85.0]
  Systolic Month 24: number analyzed (Participants) | 23 | 24
  Systolic Month 24 | 130.0 [122.0 to 142.0] | 130.0 [121.5 to 139.0]

25. Secondary Outcome: Mean Changes From Baseline Values for Blood Pressure
Description: Mean changes from baseline values for SBP and DBP at 6, 12 and 24 months post-transplant
Time Frame: Up to 24 Months
Population: ITT Population
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 26 | 32
mmHg
  Diastolic Month 6: number analyzed (Participants) | 24 | 28
  Diastolic Month 6 | 1.0 [-4.7 to 6.7] | 4.8 [-1.2 to 10.8]
  Systolic Month 6: number analyzed (Participants) | 24 | 28
  Systolic Month 6 | -4.0 [-13.9 to 5.9] | -0.7 [-10.0 to 8.7]
  Diastolic Month 12: number analyzed (Participants) | 24 | 27
  Diastolic Month 12 | 2.3 [-4.0 to 8.6] | 5.4 [-1.0 to 11.7]
  Systolic Month 12: number analyzed (Participants) | 24 | 27
  Systolic Month 12 | -1.1 [-9.6 to 7.4] | -3.2 [-14.7 to 8.3]
  Diastolic Month 24: number analyzed (Participants) | 23 | 24
  Diastolic Month 24 | 0.9 [-5.5 to 7.3] | 2.1 [-3.9 to 8.1]
  Systolic Month 24: number analyzed (Participants) | 23 | 24
  Systolic Month 24 | -2.3 [-12.2 to 7.6] | -4.2 [-14.4 to 6.0]

26. Secondary Outcome: Absolute Values of Fasting Lipid Values: Mean
Description: Absolute (mean and median) values at 3, 6, 12 and 24 months post-transplant for the following:
  Serum total cholesterol (TC) Serum high density lipoprotein (HDL) cholesterol Serum low density lipoprotein (LDL) cholesterol Serum triglycerides (TG)
Time Frame: Up to 24 Months
Population: ITT Population
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 26 | 32
mg/dL
  TC Month 3: number analyzed (Participants) | 18 | 23
  TC Month 3 | 181.2 [157.8 to 204.7] | 174.4 [154.8 to 194.1]
  TC Month 6: number analyzed (Participants) | 20 | 25
  TC Month 6 | 197.7 [177.9 to 217.4] | 175 [158.8 to 191.6]
  TC Month 12: number analyzed (Participants) | 23 | 24
  TC Month 12 | 189.0 [171.7 to 206.3] | 169.9 [153.8 to 186.0]
  TC Month 24: number analyzed (Participants) | 17 | 19
  TC Month 24 | 193.2 [172.1 to 214.2] | 168.2 [152.9 to 183.4]
  HDL Month 3: number analyzed (Participants) | 18 | 23
  HDL Month 3 | 50.6 [43.5 to 57.6] | 50.4 [43.9 to 56.9]
  HDL Month 6: number analyzed (Participants) | 20 | 25
  HDL Month 6 | 46.4 [41.3 to 51.5] | 53.9 [45.9 to 61.8]
  HDL Month 12: number analyzed (Participants) | 22 | 24
  HDL Month 12 | 49.4 [44.0 to 54.8] | 49.6 [42.5 to 56.6]
  HDL Month 24: number analyzed (Participants) | 17 | 19
  HDL Month 24 | 50.1 [44.7 to 55.5] | 51.3 [43.0 to 59.6]
  LDL Month 3: number analyzed (Participants) | 17 | 23
  LDL Month 3 | 96.9 [77.9 to 115.9] | 96.5 [80.3 to 112.6]
  LDL Month 6: number analyzed (Participants) | 20 | 25
  LDL Month 6 | 115.2 [98.1 to 132.3] | 93.7 [79.2 to 108.2]
  LDL Month 12: number analyzed (Participants) | 22 | 24
  LDL Month 12 | 107.5 [92.8 to 122.2] | 88.0 [74.3 to 101.8]
  LDL Month 24: number analyzed (Participants) | 14 | 18
  LDL Month 24 | 97.9 [81.6 to 114.2] | 91.5 [75.4 to 107.6]
  TG Month 3: number analyzed (Participants) | 18 | 23
  TG Month 3 | 171.6 [118.1 to 225.0] | 137.8 [106.6 to 168.9]
  TG Month 6: number analyzed (Participants) | 20 | 25
  TG Month 6 | 180.0 [140.2 to 219.7] | 138.3 [108.0 to 168.5]
  TG Month 12: number analyzed (Participants) | 23 | 24
  TG Month 12 | 162.4 [132.2 to 192.6] | 161.3 [126.4 to 196.1]
  TG Month 24: number analyzed (Participants) | 17 | 19
  TG Month 24 | 263.4 [131.2 to 395.5] | 145.0 [99.8 to 190.2]

27. Secondary Outcome: Absolute Values of Fasting Lipid Values: Median
Description: as for outcome 26
Time Frame: Up to 24 Months
Population: ITT Population
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 26 | 32
mg/dL
  TC Month 3: number analyzed (Participants) | 18 | 23
  TC Month 3 | 167.0 [160.0 to 213.0] | 173.0 [146.0 to 197.0]
  TC Month 6: number analyzed (Participants) | 20 | 25
  TC Month 6 | 187.0 [170.5 to 226.5] | 178.0 [146.0 to 199.0]
  TC Month 12: number analyzed (Participants) | 23 | 24
  TC Month 12 | 184.0 [166.0 to 213.0] | 171.5 [146.5 to 193.5]
  TC Month 24: number analyzed (Participants) | 17 | 19
  TC Month 24 | 193.0 [166.0 to 206.0] | 166.0 [137.0 to 201.0]
  HDL Month 3: number analyzed (Participants) | 18 | 23
  HDL Month 3 | 45.0 [39.0 to 62.0] | 49.0 [38.0 to 63.0]
  HDL Month 6: number analyzed (Participants) | 20 | 25
  HDL Month 6 | 45.5 [39.0 to 51.0] | 49.0 [37.0 to 68.0]
  HDL Month 12: number analyzed (Participants) | 22 | 24
  HDL Month 12 | 50.0 [40.0 to 58.0] | 47.0 [37.0 to 61.0]
  HDL Month 24: number analyzed (Participants) | 17 | 19
  HDL Month 24 | 49.0 [43.0 to 58.0] | 49.0 [35.0 to 71.0]
  LDL Month 3: number analyzed (Participants) | 17 | 23
  LDL Month 3 | 89.0 [74.0 to 127.0] | 95.0 [75.0 to 116.0]
  LDL Month 6: number analyzed (Participants) | 20 | 25
  LDL Month 6 | 99.5 [85.5 to 143.0] | 100.0 [66.0 to 115.0]
  LDL Month 12: number analyzed (Participants) | 22 | 24
  LDL Month 12 | 104.0 [85.0 to 128.0] | 91.5 [65.0 to 109.0]
  LDL Month 24: number analyzed (Participants) | 14 | 18
  LDL Month 24 | 103.5 [74.0 to 121.0] | 86.0 [70.0 to 119.0]
  TG Month 3: number analyzed (Participants) | 18 | 23
  TG Month 3 | 147.0 [107.0 to 195.0] | 128.0 [81.0 to 174.0]
  TG Month 6: number analyzed (Participants) | 20 | 25
  TG Month 6 | 157.5 [113.5 to 245.5] | 126.0 [85.0 to 194.0]
  TG Month 12: number analyzed (Participants) | 23 | 24
  TG Month 12 | 154.0 [100.0 to 230.0] | 130.0 [106.0 to 202.0]
  TG Month 24: number analyzed (Participants) | 17 | 19
  TG Month 24 | 159.0 [137.0 to 284.0] | 114.0 [80.0 to 174.0]

28. Secondary Outcome: Mean Changes From Baseline Values of Lipid Values
Description: Mean changes from baseline values in the following:
  Serum total cholesterol (TC) Serum high density lipoprotein (HDL) cholesterol Serum low density lipoprotein (LDL) cholesterol Serum triglycerides (TG)
Time Frame: at months 12 and 24
Population: ITT Population
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 26 | 32
mg/dL
  TC Month 12: number analyzed (Participants) | 22 | 22
  TC Month 12 | 25.7 [3.5 to 47.9] | -2.8 [-41.5 to 35.8]
  TC Month 24: number analyzed (Participants) | 16 | 17
  TC Month 24 | 26.6 [4.0 to 49.1] | 10.0 [-9.9 to 29.9]
  HDL Month 12: number analyzed (Participants) | 21 | 22
  HDL Month 12 | 5.4 [-0.3 to 11.0] | 1.9 [-3.7 to 7.5]
  HDL Month 24: number analyzed (Participants) | 16 | 17
  HDL Month 24 | 6.2 [0.7 to 11.6] | 4.8 [-2.2 to 11.9]
  LDL Month 12: number analyzed (Participants) | 20 | 16
  LDL Month 12 | 25.7 [7.9 to 43.4] | 10.8 [-10.8 to 32.4]
  LDL Month 24: number analyzed (Participants) | 11 | 12
  LDL Month 24 | 17.4 [0.0 to 34.7] | 15.7 [-4.4 to 35.7]
  TG Month 12: number analyzed (Participants) | 20 | 18
  TG Month 12 | 3.3 [-26.0 to 32.5] | -86.1 [-288.9 to 116.7]
  TG Month 24: number analyzed (Participants) | 14 | 14
  TG Month 24 | 106.8 [-32.6 to 246.2] | -13.6 [-73.8 to 46.5]

ADVERSE EVENTS:
Time Frame: Up to 24 months after last treatment dose
Description: Because 1 participant ith BPAR had been randomized to the BELA+EVL group, but had then mistakenly been treated with TAC+MMF beginning on Day 1 and continuing through the entire 2-year study period, analysis was also performed using the modified ITT (as-treated) population, in which the participant was analyzed as having received TAC+MMF.
Groups:
- BELA+EVL: BELA + EVL
- TAC+MMF: TAC + MMF
Arm/Group | BELA+EVL | TAC+MMF
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/33
Serious Adverse Events (participants affected / at risk) | 13/25 | 20/33
Other Adverse Events (participants affected / at risk) | 25/25 | 30/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BELA+EVL (N=25) | TAC+MMF (N=33)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 4
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Arteriospasm coronary (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Abdominal adhesions (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 0
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1 | 0
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 2 | 0
Renal transplant failure (Immune system disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Gastroenteritis norovirus (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Osteomyelitis acute (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Renal graft infection (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 3 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 3
Weight decreased (Investigations) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Central nervous system vasculitis (Nervous system disorders) | 0 | 1
Cerebellar ataxia (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 2
Bladder stenosis (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Nephropathy toxic (Renal and urinary disorders) | 1 | 0
Perinephric collection (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1
Renal artery stenosis (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1
Renal tubular necrosis (Renal and urinary disorders) | 1 | 1
Ureteral necrosis (Renal and urinary disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0
Dry gangrene (Vascular disorders) | 1 | 0
Iliac artery occlusion (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BELA+EVL (N=25) | TAC+MMF (N=33)
Anaemia (Blood and lymphatic system disorders) | 4 | 5
Leukocytosis (Blood and lymphatic system disorders) | 0 | 2
Leukopenia (Blood and lymphatic system disorders) | 8 | 7
Neutropenia (Blood and lymphatic system disorders) | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 4 | 1
Palpitations (Cardiac disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 2 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 4
Abdominal pain (Gastrointestinal disorders) | 2 | 3
Abdominal pain lower (Gastrointestinal disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1
Aphthous ulcer (Gastrointestinal disorders) | 4 | 2
Constipation (Gastrointestinal disorders) | 5 | 10
Diarrhoea (Gastrointestinal disorders) | 4 | 10
Dyspepsia (Gastrointestinal disorders) | 0 | 4
Flatulence (Gastrointestinal disorders) | 1 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 5
Mouth ulceration (Gastrointestinal disorders) | 10 | 0
Nausea (Gastrointestinal disorders) | 5 | 13
Vomiting (Gastrointestinal disorders) | 5 | 7
Chest pain (General disorders) | 2 | 0
Fatigue (General disorders) | 4 | 3
Oedema peripheral (General disorders) | 5 | 5
Pyrexia (General disorders) | 2 | 3
BK virus infection (Infections and infestations) | 4 | 3
Body tinea (Infections and infestations) | 2 | 0
Bronchitis (Infections and infestations) | 2 | 0
Cytomegalovirus viraemia (Infections and infestations) | 0 | 2
Fungal infection (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 1 | 3
Nasopharyngitis (Infections and infestations) | 1 | 2
Onychomycosis (Infections and infestations) | 2 | 0
Tooth infection (Infections and infestations) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 2
Urinary tract infection (Infections and infestations) | 5 | 4
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 2 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 2
Graft complication (Injury, poisoning and procedural complications) | 2 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 3
Limb injury (Injury, poisoning and procedural complications) | 0 | 2
Procedural pain (Injury, poisoning and procedural complications) | 4 | 4
Wound (Injury, poisoning and procedural complications) | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 0
Blood bicarbonate decreased (Investigations) | 0 | 2
Blood creatinine increased (Investigations) | 1 | 2
Donor specific antibody present (Investigations) | 2 | 0
Hepatic enzyme increased (Investigations) | 2 | 0
Lymphocyte count decreased (Investigations) | 0 | 2
White blood cell count decreased (Investigations) | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 5
Fluid overload (Metabolism and nutrition disorders) | 3 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 11
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 8
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 9 | 8
Metabolic acidosis (Metabolism and nutrition disorders) | 4 | 3
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Dizziness (Nervous system disorders) | 2 | 4
Headache (Nervous system disorders) | 5 | 7
Hypoaesthesia (Nervous system disorders) | 1 | 3
Paraesthesia (Nervous system disorders) | 0 | 3
Tremor (Nervous system disorders) | 0 | 6
Anxiety (Psychiatric disorders) | 2 | 1
Insomnia (Psychiatric disorders) | 3 | 5
Dysuria (Renal and urinary disorders) | 3 | 4
Haematuria (Renal and urinary disorders) | 1 | 5
Perinephric collection (Renal and urinary disorders) | 0 | 4
Proteinuria (Renal and urinary disorders) | 4 | 2
Renal impairment (Renal and urinary disorders) | 1 | 2
Renal tubular necrosis (Renal and urinary disorders) | 1 | 3
Urinary retention (Renal and urinary disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0
Hypertension (Vascular disorders) | 6 | 8
Hypotension (Vascular disorders) | 0 | 2
Orthostatic hypotension (Vascular disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
One participant with BPAR had been randomized to the BELA+EVL group, but had then mistakenly been treated with TAC+MMF beginning on Day 1 and continuing through the entire 2-year study period. Due to this, time to CSBPAR was performed using this inaccurate population, therefore inaccurate data is not presented.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-08-14): https://cdn.clinicaltrials.gov/large-docs/39/NCT02137239/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-26): https://cdn.clinicaltrials.gov/large-docs/39/NCT02137239/SAP_001.pdf